CLINICAL TRIAL: NCT06905535
Title: The Effect of Carotid Corrected Blood Flow Time Measured in the Left Lateral Tilt Position on the Prediction of Spinal Anaesthesia-induced Hypotension in Caesarean Section
Brief Title: Corrected Carotid Flow Time for Predicting Spinal Anesthesia-induced Hypotension
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Associated professor, Selcuk University
Other Study IDs: carotis flow
Record Dates: First submitted 2024-12-13; First posted 2025-04-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hypotension
Keywords: spinal anesthesia induced hypotension; carotid flow time
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Spinal anaesthesia is a standard technique frequently preferred for caesarean section. However, spinal anaesthesia-induced hypotension remains a critical problem causing undesirable maternal symptoms such as nausea, vomiting and dyspnoea and adverse consequences for umbilical acidosis and the fetus. One of the reasons aggravating hypotension is aortocaval compression of the growing uterus and consequent decrease in preload and stroke volume . Therefore, left lateral tilt position is recommended in pregnant women after the 20th gestational week to prevent supine hypotension. This position decreases uterine compression on the vena cava and increases venous return to the heart and thus stroke volume. Recently, carotid artery Doppler has been used to assess stroke volume. Many studies have shown that carotid corrected flow time increases significantly after expansion of intravascular volume in hypovolaemic patients . In one study, it was reported that the change in carotid artery blood flow time induced by passive leg raising predicts fluid sensitivity in critically ill patients. It has been reported that changes in carotid artery blood flow time against hemodynamic interventions (such as Trendelenburg position) reflect maternal hypovolemic status and distinguish hypovolemic patients with a higher risk of spinal anesthesia-related hypotension. The investigators also think that the left lateral tilt position may increase the corrected carotid flow time by affecting hemodynamics and may differentiate the patient with a high risk of hypotension.

DETAILED DESCRIPTION:
Patients undergoing elective cesarean section under spinal anesthesia will be included in the study. Carotid corrected flow time will be measured by Doppler ultrasonography in the supine and left lateral tilt (15°) positions before spinal anesthesia. Flow time will be measured using pulse Doppler waveforms in the long axis of the right common carotid artery. The measured flow time will be calculated as "corrected flow time" using the following Wodey formula; Carotid corrected flow time = measured flow time + [1.29 (Heart rate - 60)].

After standard monitoring (Electrocardiography, peripheral oxygen saturation, noninvasive blood pressure measurement), routine spinal anesthesia will be performed without any study-specific changes. The noninvasive blood pressure value measured before spinal anesthesia will be taken as the baseline value and a decrease of 20% or more in this value or a decrease in systolic blood pressure below 100 mmHg will be considered as "spinal anesthesia induced hypotension". Patients will be divided into those who develop spinal anesthesia-induced hypotension and those who do not develop spinal anesthesia-induced hypotension after spinal anesthesia and carotid corrected flow times will be compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnancy
* physical status II of American Society of Anesthesiologists

Exclusion Criteria:

* emergency cesarean section,
* cesarean under general anesthesia
* gestational Diabetes Mellitus
* gestational Hypertension
* preeclampsia,
* cardiovascular disease
* cerebrovascular disease
* chronic kidney disease disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing cesarean section in Selcuk University Faculty of Medicine Hospital Gynecology Operating Room
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
predictive value of the carotid flow time alteration | 10-15 minute
  rate of prediction